CLINICAL TRIAL: NCT06322147
Title: Doublet or Triplet Chemotherapy With Cetuximab as Conversion Therapy in RAS/BRAF Wild Type Unresectable Liver Metastasis Right-sided Colon Cancer With Curative Intent：Multi-center, Ambispective Observational Trial
Brief Title: Chemotherapy With Cetuximab as Conversion Therapy in RAS/BRAF WT Unresectable Liver Metastasis Right-sided Colon Cancer
Status: Recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: KYLL-202304-31
Record Dates: First submitted 2024-03-06; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-02

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Doublet or triplet chemotherapy combined with cetuximab
  Interventions: Drug: Doublet or triplet chemotherapy combined with cetuximab

INTERVENTIONS:
Drug: Doublet or triplet chemotherapy combined with cetuximab — chemotherapy+cetuximab combination therapy，chemotherapy regimens include FOLFOX, FOLFIRI, XELOX, or mFOLFOXIRI.
  Cetuximab first dose 400 mg/m2, followed by cetuximab 250 mg/m2 every 2 weeks;
  mFOLFOX6: oxaliplatin 85 mg/m2 (day 1), 5-FU 400 mg/m2 (day 1), LV 400 mg/m2 (day 1), and 5-FU 2400 mg/m2 CIV (46 h) for up to 12 cycles;
  XELOX (biweekly): oxaliplatin 85 mg/m2 (day 1), capecitabine 1000 mg/m2, bid, d1-10;
  FOLFIRI: irinotecan 180 mg/m2 (day 1), 5-FU 400 mg/m2 (day 1), LV 400 mg/m2 (day 1), and 5-FU 2400 mg/m2 CIV (46 h), Up to 12 cycles;
  mFOLFOXIRI: oxaliplatin 85 mg/m2 (day 1), irinotecan 150 mg/m2 (day 1), 5-FU 400 mg/m2 (day 1), LV 400 mg/m2 (day 1) and 5-FU 2400 mg/m2 CIV (46 h).

SUMMARY:
This study was designed as multi-center, ambispective observational trial to evaluate the efficacy and safety of addition of cetuximab to doublet or triplet chemotherapy as conversion therapy in right-sided BRAF/RAS wild-type CRLM with curative intent. The primary endpoint was radical resection rate (R0). The secondary endpoint was response rate, rate of NED, depth of remission, early tumor shrinkage, progression free survival and safety.

DETAILED DESCRIPTION:
Patients with colorectal liver-limited metastases (CLM) represent an exceptional subgroup with regards to the possible benefits of potentially curative multidisciplinary strategies, in which the upfront most active combination regimens are preferred to improve the rate of radical resection (R0) and NED (no evidence of disease). Unfortunately, Data are limited that specifically address the tumor location's impact on conversion therapy. As far as right-sided CRLM are concerned, much lower R0 after conversion therapy could be achieved when compared with left-sided CRLM. Furthermore, great controversies remain about the optimal conversion regimens in right-sided CRLM and the potential roles of anti-EGFR with regards to the different recommendations from NCCN, ESMO and CSCO guidelines. Chemotherapy plus cetuximab have the advantages in terms of response rate, early tumor shrinkage and depth of response, thus it is still of great value to explore the roles of cetuximab plus chemotherapy as conversion strategy in the right-sided RAS/BRAF wild type and MSS CRLM in the real world scenario.

This study was designed as multi-center, ambispective observational trial to evaluate the efficacy and safety of addition of cetuximab to doublet or triplet chemotherapy as conversion therapy in right-sided BRAF/RAS wild-type CRLM with curative intent. The primary endpoint was radical resection rate (R0). The secondary endpoint was response rate, rate of NED, depth of remission, early tumor shrinkage, progression free survival and safety.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained before any study specific procedures. Subjects must be able to understand and willing to sign a written informed consent;
* Male or female subjects > 18 years < 75 of age;
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 ;
* Life expectancy of more than 3 months;
* Patients with pathologically confirmed metastatic colorectal liver metastases with molecular testing RAS/BRAF wild-type, MSS;
* At least one measurable lesion in liver metastases according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1;
* No previous any systemic anticancer therapy; if received primary tumor surgery and postoperative adjuvant chemotherapy, more than 6 months from the end of the last chemotherapy;
* Liver metastases are initially unresectable, but can have the opportunity to achieve complete resection or NED status with conversion therapy;
* Patients have adequate bone marrow, hepatic and renal function;

Exclusion Criteria:

* Any evidence of extra-hepatic metastases, lymph node (including portal lymph nodes) metastases and primary tumor recurrence.
* The primary tumor cannot be completely resected;
* If the possibility of R0 transformation is achieved, the patient refuses surgery due to non-medical factors.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: RAS/BRAF wild type unresectable liver metastasis right-sided colon cancer
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | 1 year
  R0 resection rate upon conversion treatment with chemotherapy plus cetuximab

SECONDARY OUTCOMES:
Objective response rate | 1 year
  CR + PR rate according to RECIST
Reported adverse events | 1 year
  Number of patients with adverse events and severity according to NCI CTC 4.0
Progression free survival | 2 year
  Time from date of randomization until the date of first documented progression or date of death from any cause, whichever came first.
no evidence of disease | 1 year
  the percentage of patients who had a curative liver treatment following protocol treatment
depth of response | 1 year
  DOR means that the period from the day when either CR or PR is first confirmed until the day of documented PD or the day of death due to all causes, whichever occurs earlier.
Early Tumor Shrinkage | 1 year
  Early tumor shrinkage assessed by Response rate at week 8

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided